CLINICAL TRIAL: NCT06684951
Title: Study the Effects of Intrauterine Flushing With Low Dose Human Chorionic Gonadotropin on Ultrasound Parameter and Immunological Marker of Endometrial Receptivity of Infertile Female Undergoing ICSI Cycle
Brief Title: Effects of Intrauterine Flushing With Human Chorionic Gonadotropin on ICSI Outcome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Omayma Ismail Khalaf (Other)
Responsible Party: Sponsor-Investigator, Omayma Ismail Khalaf, principal investigator, Al-Nahrain University
Organization: Al-Nahrain University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0701-PF-2022O10
Record Dates: First submitted 2024-08-20; First posted 2024-11-12 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Female Infertility
Keywords: Implantation; Infertility; Human Chorionic Gonadotropin
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group A (Active Comparator): Intrauterine infusion of 700IU of human chorionic gonadotropin once immediately after ova pickup
  Interventions: Drug: hCG
- Group B (Active Comparator): Intrauterine infusion of 500IU of human chorionic gonadotropin once immediately after ova pickup
  Interventions: Drug: hCG
- group C (No Intervention): patient not receive any treatement

INTERVENTIONS:
Drug: hCG — observe hCG effect on endometrial receptivity
  Arms: Group A; Group B

SUMMARY:
a number of infertile women who were prepared for ICSI and immediately post ova pick up intrauterine flushing with human chorionic gonadotropin was done to study the effect of this drug on ICSI outcome and ultrasound parameter.

DETAILED DESCRIPTION:
Ninety infertile women included. Written informed consent was obtained before being included in the study. Three groups of patients according to type of intervention. Assessment of plasma hormone level was done for all. The quantification of serum TNF and IL-10 levels was conducted through the application of the enzyme-linked immunosorbent assay (ELISA) methodology at a privately-owned laboratory.

ELIGIBILITY:
Inclusion Criteria:

1. The patient's consent to participate in the research study is crucial for data collection and analysis.
2. Each pair of individuals undergoing IVF/ICSI procedures typically possess grade 1 (G1) embryos during the embryo transfer process.
3. The age range of the female participants varied from 18 to 40 years.
4. Infertility arising from female factors, including issues like blocked fallopian tubes, lack of ovulation, and unexplained fertility challenges, was examined.
5. Male-related factors contributing to infertility were also taken into consideration.
6. The procedure involved the transfer of grade one embryos during a fresh cycle.

Exclusion Criteria:

Endometrioses, whether clinically suspected or discovered during laparoscopy, are of interest.

2. Instances of congenital abnormalities in the reproductive system are being examined.

3. Individuals above the age of forty are under consideration. 4. Individuals who do not possess G1 embryos are also included. 5. Patients with chronic systemic conditions (such as diabetes, hematologic disorders, hypertension, autoimmune disorders of the connective tissue, asthma, thyroid disorders) are a part of the study.

6. The presence of empty follicles is noted in stimulated cycles where no oocytes were obtained during the aspiration procedure.

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — intertile female age (18-40), no history of endocrinological disease
Enrollment: 90 (Actual)
Dates: Start 2022-10-23 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manal T Al-Obaidi, phD., Study Director — High Institute for Infertility Diagnosis and Reproductive Technique
Locations (1):
- High Institute for Infertility Diagnosis and Assisted Reproductive Technology, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on patients whom attended the out patient clinic of the High Institute for Infertility Diagnosis and Assisted reproductive technique/ Al Nahrain university, between October 2022 and January 2024.
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 30 | 30 | 30
Completed | 30 | 30 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 30 | 30 | 30 | 90
Age, Customized [Count of Participants; unit: Participants]
  age of participants (years): Age < 25 | 5 | 4 | 4 | 13
  age of participants (years): 25-34 | 17 | 21 | 18 | 56
  age of participants (years): ≥ 35 | 8 | 5 | 8 | 21
Sex/Gender, Customized [Count of Participants; unit: Participants] — all participants were infertile female attended out patient clinic for high institute for infertility diagnosis and assisted repr0ductive technique
  Participants
    female participant | 30 | 30 | 30 | 90
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — aii patients enrolled in the study collected from high institute for infertility diagnosis and assisted reproductive technique / Al Nahrain university
  Participants
    Iraq | 30 | 30 | 30 | 90
Body mass index (BMI) Kg/m^2 [Count of Participants; unit: Participants]
  Normal BMI | 4 | 9 | 5 | 18
  over weight | 20 | 13 | 18 | 51
  obese | 6 | 8 | 7 | 21
Type of infertility (primary/secondary) [Count of Participants; unit: Participants]
  primary | 26 | 23 | 28 | 77
  secondary | 4 | 7 | 2 | 13
Cause of infertility [Count of Participants; unit: Participants]
  male factor | 22 | 23 | 19 | 64
  female factor | 1 | 4 | 6 | 11
  Combined | 2 | 2 | 2 | 6
  Unexplained | 5 | 1 | 3 | 9
Duration of infertility [Count of Participants; unit: Participants]
  < 5 years | 8 | 9 | 9 | 26
  5 - 9 years | 9 | 11 | 13 | 33
  ≥ 10 years | 13 | 10 | 8 | 31

OUTCOME MEASURES:

1. Primary Outcome: Serum Level of TNF-alfa,IL-10, for All Participants in Three Study Group at Day of Ova Pickup Compared to That at Day of Embryo Transfer
Description: All participants in the study had a blood sample taken on the day of ovum retrieval (within 10 minute after ova pickup) for the purpose of measuring the level of interleukin-10 and TNF-alfa in the blood, and a second sample was taken on the day of embryo transfer (ten minute before embryo transfer) to asses both marker,
Time Frame: at day of ova pickup a blood sample aspirated, and on day of embryo transfer about 3-5 days post ova pickup blood sample taken within ten minute before embryo transfer to asses serum level of TNF-alfa and IL-10 for all participent
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Group A: Intrauterine infusion of 700IU of human chorionic gonadotropin once immediately after ova pickup
  hCG: observe hCG effect on endometrial receptivity and biochemical marker including TNF-alfa and IL-10
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 30 | 30 | 30
pg/ml
  serum level of TNF-alfa at day of ova pickup | 43.56 (12.6) | 41.59 (8.4) | 40.94 (14.4)
  TNF-alfa day of embryo transfer | 30.33 (5.7) | 38.06 (10.6) | 42.3 (18.7)
  IL-10 day of pickup | 25.26 (10.9) | 27.08 (4.9) | 25.57 (8.3)
  IL-10 day of embryo transfer | 25.21 (14.5) | 23.4 (5.6) | 25.51 (12.8)

2. Primary Outcome: Ultrasound Parameter (RI,PI)
Description: assessment of sub-endometrial blood flow indicis immediately within 10 minute post ova pickup and second exam within ten minute before embryo transfer day which is within 3-5 days of ova pickup there are no maximum or minimum value for the parameter to be measured and lower value is better these measure was performed by using ultrasound device
Time Frame: Within 10 minutes after ova pickup, ten minute before embryo transfer using ultrasound device
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 30 | 30 | 30
index
  Resistance index day of pickup | 0.49 (0.06) | 0.51 (0.08) | 0.5 (0.05)
  Resistance index day of transfer | 0.42 (0.07) | 0.48 (0.1) | 0.5 (0.07)
  Pulsatile index day of pickup | 0.8 (0.14) | 0.85 (0.22) | 0.79 (0.16)
  Pulsatile index day of transfer | 0.64 (0.21) | 0.82 (0.25) | 0.78 (0.13)

3. Primary Outcome: Systole Flow/ Diastole Flow
Description: ultrasound parameter to asses endometrial receptivity by measuring sub-endometrial flow systole / diastole ratio
Time Frame: within ten minute post ova pickup and ten minute prior to embryo transfer which is done within 3-5 days post ova pickup
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 30 | 30 | 30
ratio
  systole/ diastole ratio day of pickup | 2.05 (0.3) | 2.3 (0.5) | 2.01 (0.3)
  systole/diastole ratio day of transfer | 1.87 (0.3) | 2.21 (0.8) | 1.92 (0.3)

4. Primary Outcome: TNF-alfa/IL-10 Ratio
Description: ratio of serum level of TNA-alfa /IL-10 at time of ova pickup and at day of embryo transfer
Time Frame: within ten minute post ova pickup and ten minute prior to embryo transfer which is done within 3-5 days post ova pickup
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 30 | 30 | 30
ratio
  TNF/IL-10 ratio at day of ova pickup | 1.89 (0.46) | 1.56 (0.33) | 1.71 (0.47)
  TNF/IL-10 ratio at day of embryo transfer | 1.38 (0.32) | 1.66 (0.38) | 1.86 (1.1)

5. Secondary Outcome: Intra Cytoplasmic Sperm Injection Outcome
Description: Number of patients who get pregnant after ICSI in each study group
Time Frame: 14 days after embryo transfer beta-hCG titer performed to asses pregnancy
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 30 | 30 | 30
Participants
  pregnant women | 16 | 12 | 8
  non-pregnant women | 14 | 18 | 22

ADVERSE EVENTS:
Time Frame: 1 year
Description: information about adverse event effect performed using questionnaire, regular laboratory testing and the intervention is by using intrauterine infusion of low dose of drug which nearly carry no risk to the patients
Arm/Group | Group A | Group B | Group C
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-10-16): https://cdn.clinicaltrials.gov/large-docs/51/NCT06684951/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-16): https://cdn.clinicaltrials.gov/large-docs/51/NCT06684951/SAP_001.pdf
  • Informed Consent Form (2024-10-16): https://cdn.clinicaltrials.gov/large-docs/51/NCT06684951/ICF_002.pdf